CLINICAL TRIAL: NCT04988477
Title: Implementation of Cessation Treatment in Community Based Mental Health Centers
Brief Title: Proactive Outreach for Smoking Treatment
Acronym: POST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sandra Japuntich (Other)
Collaborators: Brown University (Other); University of Minnesota (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Sandra Japuntich, Sandra Japuntich, Ph.D., L.P., Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-4723; 5R34DA046078 (NIH)
Record Dates: First submitted 2021-07-23; First posted 2021-08-03 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-05

CONDITIONS: Smoking, Tobacco; Mental Illness
Keywords: smoking; Chronic care model; Serious mental illness; implementation science
MeSH Terms: conditions — Tobacco Smoking; Mental Disorders; Smoking

STUDY DESIGN:
Intervention Model Description: Study 1 is a key informant interview study. Study 2 is a pre-post study. Study 3: is a pre-post study with multiple baselines to account for change over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study 3 (Experimental): Quarterly brief provider interventions about tobacco and 3 quarterly proactive outreach calls to connect patients to telephone cessation counseling and facilitate obtaining cessation medication.
  Interventions: Behavioral: Study 3: Chronic care management
- Study 2 (Experimental): In this study, participants received brief provider interventions about tobacco and a single outreach call to connect them to telephone cessation counseling and facilitate obtaining cessation medication.
  Interventions: Behavioral: Study 2: Pilot trial
- Study 1 (No Intervention): Patients, providers and leaders at community mental health centers were interviewed about intervention feasibility and acceptability

INTERVENTIONS:
Behavioral: Study 3: Chronic care management — Quarterly brief provider intervention (the 5As) and 3 quarterly outreach calls over 9 months.
  Arms: Study 3
Behavioral: Study 2: Pilot trial — Providers trained in brief provider intervention and 1 outreach call over 3 months.
  Arms: Study 2

SUMMARY:
Tobacco use disorder is a chronic disease. This is particularly true for people living with mental illness, who are more likely to smoke and make more unsuccessful quit attempts than those without. The current study is designed to test a package of two chronic disease management strategies to treatment tobacco in community mental health centers: regular provider interventions during routine mental healthcare visits, and proactive outreach by community mental health center staff to offer connections to tobacco cessation treatment. In study 1 we will interview patients, providers and leaders across wo community healthcare systems, in study 2 we will pilot test the package of interventions in 25 patients at a community mental health center for feasibility and acceptability. in Study 3, 50 patients at a community mental health center will receive provider intervention at their regular visits as well as 3 outreach calls over 9 months from trained staff to offer to connect them with stop smoking treatment. The investigators will measure the effect of these interventions on tobacco use over the next year.

DETAILED DESCRIPTION:
BACKGROUND: The US Public Health Service (USPHS) designated tobacco dependence as a chronic disease. This is especially true for smokers with serious mental illness (SMI) who make more cessation attempts and are less successful sustaining long-term abstinence than the general population. There is a significant health disparity wherein individuals with SMI have a higher tobacco use prevalence and a greater risk for tobacco-related mortality than the general population. Chronic care models suggest chronic disease management requires a multidisciplinary care team to assess tobacco use, administer treatment, support patient self-management, and monitor progress. Proactive telephone outreach to smokers and brief provider interventions are two effective chronic disease management strategies. Community based mental health centers (CMHCs) are a primary treatment access point for many smokers with SMI. However, rates of intervention with smoking by CMHC providers are low. In order to implement the chronic care model for tobacco dependence for CMHCs, comprehensive implementation strategies are needed. OBJECTIVE: to conduct a feasibility pilot trial to adapt an implementation strategy developed by the SAMHSA-funded network of Addiction Technology Transfer Centers (ATTCs) to integrate a proactive, chronic care model of tobacco cessation treatment into CMHCs. AIM: To conduct a pilot trial to assess the feasibility, acceptability and initial effectiveness of the implementation strategy. DESIGN: The investigators will conduct 3 studies. The first study will include qualitative interviews of 29 individuals including patients, providers and leaders. Study 2 will be a pilot test of the study intervention. 25 patients will receive the intervention for 3 months the primary outcome is feasibility and acceptability as measured 3 months post intervention. Study 3 is a pilot hybrid type 2 implementation-effectiveness trial in 3 CMHCs (N=50 patients; 96-130 providers). The investigators will conduct 2 baseline assessments (3 months apart) and outcomes will be assessed at 3, 6, and 12-months post implementation.

Outcomes include feasibility, acceptability, effectiveness of the implementation strategy on tobacco cessation treatment utilization (counseling and medication) and patient effectiveness on tobacco cessation (CO confirmed 7-day point prevalence abstinence). SIGNIFICANCE: An effective implementation strategy for tobacco cessation treatment in CMHCs, a widespread model of care delivery, would have enormous public health impact.

ELIGIBILITY:
Inclusion Criteria:

* daily cigarettes smokers (smoking >25 days/month)
* English speaking
* patient in one of the two community mental health center study sites.

Exclusion Criteria:

* cognitive impairment
* judged by community mental health center staff as unable to participate in research
* no access to a telephone
* no mailing address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin Healthcare Research Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Within 18 months of study completion, we will make completely de-identified data (i.e., data that has been cleaned of all 18 types of HIPAA identifiers) datasets available to interested investigators who submit a written request to the PI. The only contingency on the use of the data will be that ethical guidelines be followed (e.g., only individuals who have completed a research ethics training course will have access to the data, the data will be stored securely).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 18 months after collection of primary outcome data for 5 years post data collection.
Access Criteria: research ethics training

RESULTS

PARTICIPANT FLOW:
Groups:
- Study 3: This is a single arm pre-post trial.
  Quarterly brief provider interventions about tobacco and 3 quarterly proactive outreach calls to connect patients to telephone cessation counseling and facilitate obtaining cessation medication.
  Chronic care management: Quarterly brief provider intervention (the 5As) and 3 quarterly outreach calls over 3 months.
- Study 1: Single Interview regarding feasibility and acceptability of delivering chronic care management for smoking cessation in community mental health centers
- Study 2: Quarterly brief provider interventions and a single proactive outreach call to connect patients to telephone cessation counseling and facilitate obtaining cessation medication.
  Chronic care management: brief provider intervention (the 5As) quarterly over 3 months and one outreach call over 3 months.
Period: Overall Study
Arm/Group | Study 3 | Study 1 | Study 2
Started | 49 | 25 | 20
Completed | 41 | 23 | 20
Not Completed | 8 | 2 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a single arm, pre-post study. Thus, we report the data for the full sample.
Groups:
- Study 3: Quarterly brief provider interventions about tobacco and 3 quarterly proactive outreach calls to connect patients to telephone cessation counseling and facilitate obtaining cessation medication.
  Chronic care management: Quarterly brief provider intervention (the 5As) and 3 quarterly outreach calls over 3 months.
- Total: Total of all reporting groups
Arm/Group | Study 3 | Study 2 | Study 1 | Total
Number analyzed (Participants) | 49 | 25 | 20 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographics were not collected in Study 1; age only collected for 48 patients in study 3
  years
    number analyzed (Participants) | 48 | 25 | 0 | 73
    (all) | 41.23 (11.88) | 48.64 (12.14) |  | 43.93 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographics were not collected in study 1
  Participants
    number analyzed (Participants) | 49 | 25 | 0 | 74
    Female | 32 | 17 |  | 49
    Male | 17 | 8 |  | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographics were not collected in Study 1
  Participants
    number analyzed (Participants) | 49 | 25 | 0 | 74
    Hispanic or Latino | 0 | 0 |  | 0
    Not Hispanic or Latino | 49 | 25 |  | 74
    Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: demographics were not collected in Study 1
  Participants
    number analyzed (Participants) | 49 | 25 | 0 | 74
    American Indian or Alaska Native | 1 | 2 |  | 3
    Asian | 0 | 0 |  | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
    Black or African American | 3 | 1 |  | 4
    White | 44 | 22 |  | 66
    More than one race | 1 | 0 |  | 1
    Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 25 | 20 | 94
cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] — Cigarettes per day was not collected in Study 1 Population: Cigarettes per day was not collected in Study 1
  cigarettes per day
    number analyzed (Participants) | 49 | 25 | 0 | 74
    (all) | 15.35 (8.97) | 16.67 (10.07) |  | 15.92 (9.30)

OUTCOME MEASURES:

1. Primary Outcome: Study 3: Smoking Abstinence
Description: number of participants who reported 7-day point prevalence smoking abstinence (no smoking past 7 days) and a expired air CO value of <6ppm in study 3 only
Time Frame: 1 year post baseline
Population: Participants who completed baseline data and were alive at follow-up (1 participant died and so data was not analyzed)
Measure: Count of Participants; unit: Participants
Arm/Group | Study 3
Number analyzed (Participants) | 48
Participants | 3

2. Primary Outcome: Study 1: Perceived Feasibility of Intervention
Description: Number of participants who reported the proposed intervention was feasible
Time Frame: interview (up to 30 minutes at study visit)
Population: Interview participants including patients, providers, and leaders at community mental health centers
Measure: Count of Participants; unit: Participants
Groups:
- Study 1: Participants were interviewed about current smoking cessation practices in their organization and feasibility and acceptability of planned study interventions
Arm/Group | Study 1
Number analyzed (Participants) | 20
Participants | 17

3. Primary Outcome: Study 1: Perceived Acceptability of Intervention
Description: number of participants who agreed the proposed intervention was acceptable.
Time Frame: interview (up to 30 minutes at study visit)
Population: patients, providers, and leaders at a community mental healthcare center
Measure: Count of Participants; unit: Participants
Arm/Group | Study 1
Number analyzed (Participants) | 20
Participants | 18

4. Primary Outcome: Studies 2 & 3: Feasibility of Recruitment
Description: Number of participants recruited (goal for study 2=25; goal for study 3=50)
Time Frame: baseline
Population: patients in a community mental healthcare center who smoke cigarettes
Measure: Count of Participants; unit: Participants
Groups:
- Study 2: In this study, participants received brief provider interventions about tobacco and a single outreach call to connect them to telephone cessation counseling and facilitate obtaining cessation medication.
  Chronic care management: Quarterly brief provider intervention (the 5As) and 3 quarterly outreach calls over 3 months.
Arm/Group | Study 2 | Study 3
Number analyzed (Participants) | 25 | 49
Participants | 25 | 49

5. Primary Outcome: Studies 2 & 3: Feasibility of Retention
Description: % of participants completing follow-up in studies 2 & 3
Time Frame: 3 months post enrollment
Population: This measure was the primary outcome of the chronic care for tobacco use (study 3) and the pilot trial (study 2) only. The recruitment target for study 2 was 25, the recruitment target for study 3 was 50.
Measure: Count of Participants; unit: Participants
Arm/Group | Study 3 | Study 2
Number analyzed (Participants) | 49 | 23
Participants | 41 | 23

6. Primary Outcome: Study 2: Perceived Acceptability of Intervention
Description: Number of participants who perceived that the intervention was acceptable drawn from qualitative reports of intervention acceptability from selected patients (N=5) and providers and leaders (N=4)
Time Frame: 3 months post enrollment
Population: Patients and providers from a community mental health center who participated in the study
Measure: Count of Participants; unit: Participants
Groups:
- Study 2: Participants received 1 outreach call from an interventionist with the offer to connect them to smoking cessation treatment. At the end of the study we conducted interviews on study acceptability.
Arm/Group | Study 2
Number analyzed (Participants) | 9
Participants | 8

7. Secondary Outcome: Study 3: Smoking Abstinence
Description: 30 day prolonged abstinence (no smoking past 30 days prior to 1 year follow-up)
Time Frame: 1 year post baseline
Population: Participants who completed baseline and were alive at the 12 month follow-up (1 participant died during the follow up period and so the did not contribute outcome data).
Measure: Count of Participants; unit: Participants
Arm/Group | Study 3
Number analyzed (Participants) | 48
Participants | 3

8. Secondary Outcome: Study 3: Quit Attempts
Description: Number of 24 hour intentional quit attempts
Time Frame: 1 year post-baseline
Population: Participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | Study 3
Number analyzed (Participants) | 49
quit attempts | 3.07 (4.46)

9. Secondary Outcome: Study 3: Cigarettes Per Day
Description: number of cigarettes smoked per day in study 3
Time Frame: 12 months post baseline
Population: participants who were alive at the 12 month follow-up (1 person died and so their data was not used)
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Study 3
Number analyzed (Participants) | 48
cigarettes per day | 10.56 (12.02)

ADVERSE EVENTS:
Time Frame: 15 months
Description: Adverse events were not systematically collected. However, if participants reported an adverse event or serious adverse event during follow-up phone calls it was documented. Additionally, if a participant was not available for follow-up due to a serious adverse event or death, that was recorded.
Groups:
- Study 3: Chronic care for tobacco use: Quarterly brief provider interventions about tobacco and 3 quarterly proactive outreach calls to connect patients to telephone cessation counseling and facilitate obtaining cessation medication.
  Chronic care management: Quarterly brief provider intervention (the 5As) and 3 quarterly outreach calls over 9 months.
- Study 2: Pilot trial: Provider brief provider interventions about tobacco and 1 proactive outreach calls to connect patients to telephone cessation counseling and facilitate obtaining cessation medication.
- Study 1: Interview study: patients, providers, and leaders were interviewed about study feasibility/acceptability
Arm/Group | Study 3: Chronic care for tobacco use | Study 2: Pilot trial | Study 1: Interview study
All-Cause Mortality (participants affected / at risk) | 1/49 | 0/25 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 0/49 | 0/25 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 3: Chronic care for tobacco use (N=49) | Study 2: Pilot trial (N=25) | Study 1: Interview study (N=20)
Inpatient Hospitalization (Injury, poisoning and procedural complications) | 1 (1) | NA | NA — Complications following a hernia repair

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT04988477/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT04988477/ICF_001.pdf